CLINICAL TRIAL: NCT00889343
Title: A Controlled Randomized Double-blind Multi-center Phase II Study of FOLFOX6 or FOLFIRI Combined With Sorafenib Versus Placebo in Second-line Metastatic Colorectal Carcinoma
Brief Title: Study to Evaluate the Effects of Sorafenib if Combined With Chemotherapy (FOLFOX6 or FOLFIRI) in the Second-Line Treatment of Colorectal Cancer
Acronym: FOSCO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AIO KRK 0307
Record Dates: First submitted 2009-04-17; First posted 2009-04-28 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Colorectal Neoplasms
Keywords: Second-line therapy of metastatic colorectal cancer; Sorafenib; Colorectal Neoplasms; palliative therapy; after progression of firstline therapy with an Oxaliplatin- or Irinotecan based Fluoropyrimidine containing regimen ± bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Sorafenib; Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Sorafenib; Drug: Oxaliplatin or Irinotecan; Drug: Leucovorin; Drug: 5-Fluorouracil
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Oxaliplatin or Irinotecan; Drug: Leucovorin; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: Sorafenib — 2x200 mg filmcoated tablets BID on day 2-12 of a 14-days cycle, oral
  Other Names: Nexavar
  Arms: 1
Drug: Placebo — 2 filmcoated tablets BID, day 2-12 of a 14-days cycle, oral
  Arms: 2
Drug: Oxaliplatin or Irinotecan — Oxaliplatin 100 mg/m2 intravenous infusion on day 1 of 14-days cycle, Irinotecan 180 mg/m2 intravenous infusion on day 1 of 14-days cycle
Drug: Leucovorin — 400 mg/m2 intravenous infusion on day 1 of a 14-days cycle
Drug: 5-Fluorouracil — 400 mg/m2 intravenous bolus infusion on day 1, 2400 mg/m2 46 hour intravenous infusion on day 1 to 2 of a 14-days cycle

SUMMARY:
The purpose of this study is to determine whether sorafenib in combination with chemotherapy has a positive effect on time to progression of the tumor or death for the treatment of large bowel cancer that has already progressed during a first chemotherapy.

DETAILED DESCRIPTION:
Patients with metastatic CRC who received a first-line therapy with an Oxaliplatin- or Irinotecan based Fluoropyrimidine containing regimen ± bevacizumab and had a progression subsequently, are eligible for this study. Patients will be randomized to receive chemotherapy (FOLFOX6 or FOLFIRI) + sorafenib 400 mg bid or chemotherapy + placebo. Patients who have received an Oxaliplatin based Fluoropyrimidine containing regimen in first-line will obtain FOLFIRI during this study. Patients who have received an Irinotecan based Fluoropyrimidine containing regimen in first-line will obtain FOLFOX6.

Primary objective of the study is to compare the Progression-free-survival (PFS) between patients receiving chemotherapy (FOLFOX6 or FOLFIRI) + sorafenib with chemotherapy + placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* ECOG Performance Status of 0 to 2
* Life expectancy of at least 12 weeks.
* Subjects with at least one uni-dimensional (RECIST) measurable lesion of metastatic colorectal carcinoma after first-line chemotherapy with an Oxaliplatin- or Irinotecan based Fluoropyrimidine containing regimen ± bevacizumab and had a progression subsequently. Lesions must be measured by CT-scan or MRI.
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:
* Hemoglobin > 9.0 g/dl
* Absolute neutrophil count (ANC) >1,500/mm3
* Platelet count 100,000/μl Total bilirubin < 1.5 times the upper limit of normal
* ALT and AST < 2.5 x upper limit of normal (< 5 x upper limit of normal for patients with liver involvement of their cancer)
* Alkaline phosphatase < 4 x upper limit of normal
* PT-INR/PTT < 1.5 x upper limit of normal [Patients who are being therapeutically anticoagulated with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists.]
* Serum creatinine < 1.5 x upper limit of normal
* Signed and dated informed consent before the start of specific protocol procedures

Exclusion Criteria:

* History of cardiac disease: congestive heart failure >NYHA class 2; active CAD (MI more than 6 mo prior to study entry is allowed); cardiac arrythmias requiring anti-arrythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension
* History of HIV infection or chronic hepatitis B or C
* Active clinically serious infections (> grade 2 NCI-CTC version 3.0)
* Symptomatic metastatic brain or meningeal tumors (unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry)
* Patients with seizure disorder requiring medication (such as steroids or anti-epileptics)
* History of organ allograft
* Patients with evidence or history of bleeding diathesis
* Patients undergoing renal dialysis
* Known deficit in Dihydropyrimidine Deshydrogenase (DPD)
* Contraindications for the use of atropine in patients receiving FOLFIRI
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry.
* Peripheral sensory neuropathy > CTC grade 2
* Chronic inflammatory bowel disease; ileus; genetic fructose intolerance
* Pregnant or breast-feeding patients.
* Women of childbearing potential must have a negative pregnancy test performed within 7 days before the start of treatment. Fertile women and men (<2 years after last menstruation in women) must use effective means of contraception (intrauterine contraceptive device, contraceptive implants, injectables (hormonal depot), transdermal hormonal contraception (contraceptive patch), sexual abstinence or vasectomised partner) during treatment and for at least 6 months after last administration of medication.
* Substance abuse, medical, psychological or social conditions that may interfere with the patient"s participation in the study or evaluation of the study results
* Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study 18. Patients unable to swallow oral medications.
* Any other anticancer chemotherapy or immunotherapy during the study or within 4 weeks of study entry.
* Radiotherapy during study or within 3 weeks of start of study drug. (Palliative radiotherapy will be allowed). Major surgery within 4 weeks of start of study
* Autologous bone marrow transplant or stem cell rescue within 4 months prior to study treatment
* Use of biologic response modifiers, such as G-CSF, within 3 week of study entry. [G-CSF and other hematopoietic growth factors may be used in the management of acute toxicity such as febrile neutropenia when clinically indicated or at the discretion of the investigator, however, they may not be substituted for a required dose reduction.] [Patients taking chronic erythropoietin are permitted provided no dose adjustment is undertaken within 2 months prior to the study or during the study]
* Investigational drug therapy outside of this trial during or within 4 weeks of study entry
* Prior exposure to the study drug.
* Any St. John´s wort containing remedy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2009-03; Primary Completion 2011-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To compare the PFS between patients receiving chemotherapy (FOLFOX6 or FOLFIRI) + sorafenib with chemotherapy + placebo | 6 to 12 months

SECONDARY OUTCOMES:
Disease control rate | 6 to 12 months
Overall survival | 6 to 12 months
Response rates | 6 to 12 months
Safety | signature of informed consent until 30 days after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Höhler, Prof. Dr. med., Principal Investigator
Locations (57):
- Germany (57):
  - Ostalb-Klinikum Aalen, Medizinische Klinik 1, Aalen, Baden-Wurttemberg
  - Kreiskliniken Esslingen gGmbH, Klinik Nürtingen, Medizinische Klinik I, Nürtingen, Baden-Wurttemberg
  - Gemeinschaftspraxis Onkologie Ravensburg, Ravensburg, Baden-Wurttemberg
  - Gemeinschaftspraxis Dr. med. U. Banhardt, Dr. med. T. Fietz, Singen, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Zentrum für Innere Medizin, Klinik für Innere Medizin I, Ulm, Baden-Wurttemberg
  - Medizinisches Versorgungszentrum am Siloah St. Trudpert Klinikum, Pforzheim, Baden-Würtemberg
  - Überörtliche Gemeinschaftspraxis Dres. Wilke und Wagner, Fürth, Bavaria
  - Hämatologischonkologische Schwerpunktpraxis, Herrsching am Ammersee, Bavaria
  - Hämatologie Onkologie Tagesklinik Landshut, Landshut, Bavaria
  - Hämato-Onkologische Schwerpunktpraxis Prof. Salat / Dr. Stoetzer / Prof. Hiller, München, Bavaria
  - Leopoldina-Krankenhaus, Medizinische Klinik II, Schweinfurt, Bavaria
  - Kreiskliniken Traunstein -Trostberg GmbH , Innere Medizin/ Hämatologie und Onkologie, Trostberg an der Alz, Bavaria
  - DIAKO Ev. Diakonie-Krankenhaus gGmbH, Medizinische Klinik II, Bremen, City state Bremen
  - MVZ für Innere Medizin in Hamburg Eppendorf, Hamburg, Hamburg
  - Klinikum Darmstadt, Medizinische Klinik V, Darmstadt, Hesse
  - Städtische Kliniken Frankfurt a.M. - Höchst, Klinik für Innere Medizin Abt. 3, Frankfurt a.M., Hesse
  - Vitanus GmbH, Frankfurt am Main, Hesse
  - Klinikum Fulda, Tumorklinik, Fulda, Hesse
  - Onkologische Praxisgemeinschaft Dres. Siehl, Söling und Prof. Hirschmann, Kassel, Hesse
  - Philipps-Universität, Klinikum Marburg, Klinik für Innere Medizin mit SP Hämatologie und Onkologie, Marburg, Hesse
  - Gemeinschaftspraxis für Hämatologie und Internistische Onkologie, Offenbach, Hesse
  - Lahn-Dill-Kliniken GmbH, Darmzentrum, Wetzlar, Hesse
  - MediProjekt, Gesellschaft für Medizinstatistik und Projektentwicklung, Hanover, Lower Saxony
  - Krankenhaus Siloah, Medizinische Klinik III, Hanover, Lower Saxony
  - Medizinische Hochschule Hannover, Klinik für Gastroenterologie, Hepatologie, Endokrinologie, Hanover, Lower Saxony
  - Onkologische Schwerpunktpraxis Hildesheim, Hildesheim, Lower Saxony
  - Hämatologie u. Internistische Onkologie, Lehrte, Lower Saxony
  - Hämatologisch-onkologische Schwerpunktpraxis Northeim, Northeim, Lower Saxony
  - Niels-Stensen-Kliniken, Marienhospital Osnabrück GmbH,, Osnabrück, Lower Saxony
  - Diakoniekrankenhaus Rotenburg (Wümme) gGmbH, I. Chirurgische Klinik, Rotenburg (Wümme), Lower Saxony
  - Praxisgemeinschaft Dr. Hancken und Partner, Onkologische Schwerpunktpraxis, Stade, Lower Saxony
  - Universitätsklinikum Rostock, Klinik für Innere Medizin, Rostock, Mecklenburg-Vorpommern
  - Wissenschaftskontor Nord GmbH und Co KG, Rostock, Mecklenburg-Vorpommern
  - Medizinische Universitätsklinik-Knappschaftskrankenhaus, Medizinische Klinik, Bochum, North Rhine-Westphalia
  - Gemeinschaftspraxis für Hämatologie und Onkologie am Sachsenring, Cologne, North Rhine-Westphalia
  - St. Vincenz-Krankenhaus, Medizinische Klinik I, Datteln, North Rhine-Westphalia
  - St. Antonius Hospital, Klinik für Hämatologie / Onkologie, Eschweiler, North Rhine-Westphalia
  - Hämato-Onkologisches Gemeinschaftspraxis, Essen, North Rhine-Westphalia
  - Katholisches Krankenhaus Hagen gem. GmbH, Klinik für Hämatologie und Onkologie, Hagen, North Rhine-Westphalia
  - Klinikum Leverkusen gGmbH, Medizinische Klinik III, Leverkusen, North Rhine-Westphalia
  - Gemeinschaftspraxis Hämatologie und Onkologie, Münster, North Rhine-Westphalia
  - Praxis und Tagesklinik für Internistische Onkologie und Hämatologie, Recklinghausen, North Rhine-Westphalia
  - Prosperhospital Recklinghausen, Medizinische Klinik I, Recklinghausen, North Rhine-Westphalia
  - Internistische Gemeinschaftspraxis, Witten, North Rhine-Westphalia
  - HELIOS Klinikum Wuppertal , Medizinische Klinik I, Wuppertal, North Rhine-Westphalia
  - I. Medizinische Klinik und Poliklinik der Johannes Gutenberg-Universität Mainz, Mainz, Rhineland-Palatinate
  - Klinikum Mutterhaus der Borromäerinnen gGmbH, Innere Medizin I, Trier, Rhineland-Palatinate
  - Universitätskliniken des Saarlandes, Innere Medizin I, Homburg / Saar, Saarland
  - Hämatologisch-onkologische Praxis Dr. med. Peter Schmidt, Neunkirchen, Saarland
  - Praxisgemeinschaft Dr. med. Thomas Göhler und Steffen Dörfel, Dresden, Saxony
  - Internistische Praxis & Tagesklinik, Neutstadt/Sachsen, Saxony
  - Städtisches Klinikum Dessau, Klinik für Innere Medizin, Dessau, Saxony-Anhalt
  - Onkologische Gemeinschaftspraxis, Halle, Saxony-Anhalt
  - Gemeinschaftspraxis für Hämatologie und Internistische Onkologie, Magdeburg, Saxony-Anhalt
  - Friedrich-Ebert-Krankenhaus Neumünster, Klinik für Hämatologie, Onkologie und Nephrologie, Neumünster, Schleswig-Holstein
  - eps-early phase solution GmbH, Jena, Thuringia
  - Sophien- und Hufeland-Klinikum gGmbH, Klinik für Innere Medizin II, Weimar, Thuringia

REFERENCES:
- See also: Arbeitsgemeinschaft der internistischen Onkologie — http://www.aio-portal.de